CLINICAL TRIAL: NCT06603818
Title: A Phase II Study of Immunotherapies (Tiragolumab and Atezolizumab) in Combination With Stereotactic Body Radiation Radiotherapy in Microsatellite Stable (MSS) Metastatic Colorectal Cancer (mCRC)
Brief Title: Immunotherapies in Combination With Stereotactic Body Radiation Radiotherapy in Microsatellite Stable (MSS) Metastatic Colorectal Cancer (mCRC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001589; 001589-C
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07-16

CONDITIONS: Microsatellite Stable Metastatic Colorectal Cancer; Metastatic Colorectal Cancer; Colorectal Cancer
Keywords: Stereotactic Body Radiation Radiotherapy; Immunotherapy; Radiation Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tiragolumab; atezolizumab; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Atezolizumab and tiragolumab IV every 3 weeks cycle plus SBRT on Days 1, 3, and 5 of Cycle 1
  Interventions: Biological: Tiragolumab; Biological: Atezolizumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Biological: Tiragolumab — Tiragolumab is given intravenously (IV) every 3 weeks (21-day cycles) for up to 2 years
Biological: Atezolizumab — Atezolizumab is given intravenously (IV) every 3 weeks (21-day cycles) for up to 2 years
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will occur on Days 1, 3, and 5 of Cycle 1 only

SUMMARY:
Background:

Metastatic colorectal cancer (mCRC) is cancer that has spread beyond the colon and rectum. Most people with mCRC die within 5 years. New immune-based treatments are making progress with some types of colon cancer. But these treatments do little for people with a type of cancer that is microsatellite stable (MSS). MSS is a specific cancer biomarker. Better treatments are needed.

Objective:

To test 2 drugs (tiragolumab and atezolizumab) combined with radiation therapy in people with MSS mCRC.

Eligibility:

People aged 18 years and older with MSS mCRC.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have imaging scans and a test of their heart function. They will provide a tissue sample from their tumor; if one is not already available, a new sample will be taken. Their ability to perform normal tasks will be assessed.

Tiragolumab and atezolizumab are both administered through a tube attached to a needle inserted into a vein. Participants will receive both drugs on day 1 of 3-week treatment cycles. Each study visit should last about 8 hours.

Participants will receive radiation therapy on days 1, 3, and 5 of cycle 1 only.

Blood samples and rectal swabs will be collected on day 1 of every cycle.

Imaging scans will be repeated every 9 weeks. Additional tumor samples may be taken during treatment.

Treatment will continue for up to 2 years.

Participants will have a follow-up visit 1 month after treatment ends. Follow-up visits will continue every 3 months for 1 more year.

DETAILED DESCRIPTION:
Background:

* Metastatic colorectal cancer (mCRC) is incurable for most patients and carries a poor diagnosis.
* Immune-based approaches in solid tumor malignancies have seen much progress but these have limited efficacy for microsatellite stable (MSS) mCRC.
* The Gastrointestinal Malignancies Section at NCI conducted a Pilot Study of the PD-1 Targeting Agent AMP-224 with low-dose cyclophosphamide and stereotactic body radiation therapy (SBRT) that supports potential antitumor efficacy of the combination of immunotherapy and radiation in MSS mCRC (NCT02298946).
* T cell immunoreceptor with Ig and ITIM domains (TIGIT) is an inhibitory receptor expressed in multiple cancers on tumor-infiltrating cytotoxic T cells, helper T cells, natural killer (NK) cells, and regulatory T cells. Its main ligand, CD155, is expressed on tumor-infiltrating myeloid cells and upregulated on cancer cells, contributing to local immune-surveillance suppression.
* Among inhibitory immune checkpoint molecules, a unique property of TIGIT blockade is that it enhances not only anti-tumor effector T-cell responses, but also NK-cell responses, and reduces the suppressive capacity of regulatory T cells.
* Pre-clinical studies show that the co-blockade of TIGIT and the programmed cell death protein 1 (PD-1) / programmed cell death ligand 1 (PD-L1) pathway may lead to decreased tumor volume. Notably, this has been observed in anti-PD-1 resistant tumor models.
* Preclinical and clinical evidence suggests further increased benefit to the double immune checkpoint blockade through increased expression of PD-L1 and neoantigens in response to SBRT.
* Early results from clinical trials suggest clinical activity of anti-TIGITplus anti-PD-L1 in solid tumors and the effect of combining immunotherapy with radiation in heavily pretreated MSS mCRC patients providing a proof of concept that radiation enhances immunotherapy response.
* A combination of anti-PD-L1, anti-TIGIT, and SBRT may increase CRC susceptibility to immune therapy given the promising activity of anti-TIGIT in combination with anti-PDL1 in preclinical studies of mice bearing subcutaneous CT26 colon tumors.

Primary Objectives:

* To confirm the Recommended Phase II dose (RP2D) of the combination therapy (tiragolumab and atezolizumab plus SBRT) in participants with MSS mCRC (Part A)
* To determine the proportion of participants without progression after 9 weeks of the combination therapy (tiragolumab and atezolizumab plus SBRT) in participants with MSS mCRC (Part B)

Eligibility:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1
* Histopathologic confirmation of mCRC by the NCI Laboratory of Pathology (LP)
* Disease not amenable to curative resection
* At least 1 lesion amenable to SBRT and a second lesion outside the radiation field to serve as a target lesion
* Adequate organ and marrow function

Design:

* This is a phase II, single-arm, non-randomized, trial using tiragolumab and atezolizumab in combination with SBRT.
* A maximum of 30 participants with MSS mCRC will be enrolled.
* Participants will receive atezolizumab and tiragolumab intravenously (IV) every 3 weeks (21-day cycles) with SBRT occurring on Days 1, 3, and 5 of Cycle 1 for 2 years.
* Participants will be evaluated routinely for toxicity and will have re-staging imaging every 9 weeks (every 3 cycles).
* Optional research biopsies will be done at baseline and during week 1 of cycle 2. If the participant has disease progression after cycle 3, a post-treatment biopsy may be performed.
* The proportion of participants that are progression-free at 9 weeks will be evaluated as a binary endpoint.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed colorectal cancer (CRC) by the NCI Laboratory of Pathology (LP). Note: Participants must provide tumor sample or be willing to undergo biopsy to confirm the diagnosis.
* Evidence of metastatic involvement.
* History of microsatellite stable (MSS) status.
* Age >= 18 years.
* Weight > 35 kg.
* ECOG performance status <= 1
* Must have measurable disease, per RECIST 1.1
* At least 2 lesions present, one of which must be amenable to SBRT and second lesion outside the radiation field must serve as target lesion to evaluate measurable disease.
* Must have progression of disease, been treated or intolerant to at least 2 lines of systemic standard of care treatment in the metastatic setting (e.g., fluoropyrimidine-, oxaliplatin-, or irinotecan-based therapy [unless ineligible for any of these drugs]).
* Participants with a history of RAS wild-type tumor must have progressed, been intolerant of OR refused anti-EGFR based treatment.
* Participants must have adequate organ and marrow function as defined below:

  * Leukocytes >= 3,000/microL
  * Absolute neutrophil count >= 1,500/microL
  * Lymphocyte count > 500/microL
  * Platelets >= 100,000/microL without transfusion or at least > 48 hours post-completion of blood transfusion
  * Hemoglobin >= 9 g/dL without transfusion or at least > 48 hours post-completion of blood transfusion
  * International normalized ratio <=1.5 x institutional upper limit of normal
  * (INR) and partial thromboplastin time (aPTT) (ULN) (if not receiving therapeutic anticoagulation)
  * Serum albumin > 2.5 g/dL
  * Total bilirubin <= 1.5 x ULN
  * Aspartate aminotransferase (AST) <= 2.5 x institutional ULN
  * Alanine transaminase (ALT) <= 2.5 x institutional ULN
  * Alkaline phosphatase (ALP) <= 2.5 x institutional ULN
  * Creatinine clearance calculated by Chronic Kidney Disease Epidemiology Collaboration (CKDEPI) equation >= 50 mL/min/1.73 m^2 for participants with creatinine levels >= 1.5 mg/dL
* Participants receiving therapeutic anticoagulation must be on an established, stable anticoagulation regimen prior to starting the study therapy.
* Negative human immunodeficiency virus (HIV) serological testing at screening.
* Participants seropositive for hepatitis B virus (HBV) antibody test are eligible if at screening:

  * have a negative HBV DNA test and
  * not on treatment with anti-viral therapy for HBV.
* Participants seropositive for hepatitis C virus (HCV) antibody test, are eligible if have a negative HCV RNA test at screening.
* Participants seropositive for Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test are eligible if have a negative EBV polymerase chain reaction (PCR) test at screening.
* Participants must have recovered from prior toxicity or adverse events to grade <= 2 per Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
* Women of child-bearing potential (WOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device [IUD], surgical sterilization, abstinence) at the study entry and up to 5 months after the last dose of the study drugs (restriction period).

Note: A woman is considered to be of child-bearing potential if she is postmenarchal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (i.e., removal of ovaries, fallopian tubes, and/or uterus).

* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 5 months after the last dose of the study drugs.
* Participants must be willing to co-enroll in protocol 11-C-0112, Acquisition of Blood and Tumor Tissue Samples from Patients with Gastrointestinal Cancer .
* Participants must understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Disease amenable to curative resection.
* Chemotherapy, radiation therapy, or biologic therapy within 3 weeks (or >= 5 half-lives, whichever is shorter) prior to starting the study therapy.
* Treatment with an investigational therapy within 42 days prior to starting the study therapy.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to starting the study therapy.
* History of prior treatment with TIGIT-directed treatment agents or other types of immunotherapies (e.g., prior treatment with CD137 agonists or investigational immune checkpoint blockade therapies, including anti-TIGIT, anti-PD1/anti-PDL1, anti-CTLA-4, anti-LAG3).
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor-alpha [TNF-alpha] agents) within 2 weeks prior to starting the study therapy, or anticipation of a need for systemic immunosuppressive medication during study therapy, with the following exceptions:

  --acute, low-dose systemic immunosuppressant medication (< 10 mg of prednisone daily) or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy).
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to starting the study therapy.
* Treatment with a live, attenuated vaccine within 4 weeks prior to starting the study therapy.
* Major surgery within 4 weeks prior to starting the study therapy.
* Prior allogeneic stem cell or solid organ transplantation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tiragolumab and atezolizumab or other agents used in a study or known hypersensitivity to Chinese hamster ovary cell products.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* History of central nervous system (CNS) metastasis or leptomeningeal disease.
* Current uncontrolled tumor-related pain. Participants requiring pain medication must be on a stable regimen at study entry.
* Current or history of chronic autoimmune disease or immune deficiency (e.g., Addison s disease, multiple sclerosis, Graves disease, Hashimoto s thyroiditis, rheumatoid arthritis, hypophysitis, systemic lupus erythematosus, Wegener s granulomatosis, sarcoidosis syndrome, etc.) or other connective tissue diseases except:

  * Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone;
  * Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen.
  * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all following conditions are met:

    * Rash must cover < 10% of body surface area
    * The disease is well controlled at screening and requires only low-potency topical corticosteroids
    * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet, radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within 12 months prior to starting the study therapy.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN).
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Severe infection within 4 weeks prior to starting the study therapy. This includes but is not limited to, hospitalizations for complications of infection, bacteremia, severe pneumonia, or any active infection that could impact participant safety.
* Active tuberculosis.
* History of significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to starting the study therapy, unstable arrhythmia, or unstable angina within 1 year prior to starting the study therapy.
* Prior invasive malignancy, (with the exception of non-melanomatous skin cancer) unless disease-free per standard of care for a minimum of 3 years prior to starting the study therapy.
* Women of childbearing potential must have a negative serum pregnancy test result at screening.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of investigational drugs, may affect the interpretation of the results or may render the participants at high risk of treatment complications.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Confirm the recommended phase II dose (RP2D) of the combination therapy | Start of therapy through cycle 1 day 21
  Dose-limiting toxicities (DLTs) will be collected and reported by type, grade and frequency.
Determine the proportion of participants without progression after 9 weeks of the combination therapy | After 9 weeks of treatment
  Proportion of participants attaining 9-week progression-free survival will be evaluated and reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Safety | Start of therapy through 28 days after last study treatment intervention.
  For safety, the number of adverse events by grade and type will be reported. The adverse events noted within the safety lead-in Part A will be reported separately as well as being a portion of the overall safety profile for the trial.
Tolerability | Start of therapy through 28 days after last study treatment intervention.
  The proportions of participants who tolerated 2 cycles of tiragolumab and atezolizumab in combination with SBRT. The observed proportions will be reported along with a 95% confidence interval.
Best overall response (Partial Response + Complete Response) according to RECIST v1.1 | Every 9 weeks during the study treatment and every 3 months after that until progression or 3 years after treatment initiation
  The BOR will be obtained along with a 95% confidence interval.
Progression Free Survival | Every 9 weeks during the study treatment and every 3 months after that until progression or 3 years after treatment initiation
  This secondary objective will provide the conventional PFS evaluation based on Kaplan-Meier curves reflecting censoring for participants not documented to reach this timepoint as appropriate. A 95% confidence interval for the median PFS will also be provided.
Overall Survival | Start of therapy until death or 3 years after treatment initiation
  The OS will be determined using the Kaplan-Meier method beginning at the date the treatment begins, along with a 95% confidence interval for the median OS.

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review. This study will comply with the NIH Genomic Data Sharing (GDS) Policy, which applies to all new and ongoing NIH IRP-funded research, as of January 25, 2015, that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested after the completion of the primary endpoint
Access Criteria: Data from this study may be requested by contacting the NCI Principal Investigator@@@@@@

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001589-C.html